CLINICAL TRIAL: NCT03433222
Title: EBIRE: Phase 1 Study of High Fluence LED-Red Light in Fitzpatrick Skin Types I to III
Brief Title: Phase 1 Study of HF-LED-RL in Fitzpatrick Skin Types I to III
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Collaborators: East Bay Institute for Research and Education (Other)
Responsible Party: Principal Investigator, Jared Jagdeo, MD, MS, Physician, Dermatology, VA Northern California Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-01-00804
Record Dates: First submitted 2018-02-01; First posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Skin Diseases; Keloid; Scar; Fibrosis; Hypertrophic Skin
Keywords: light emitting diode-red light; high fluence; red light; RCT
MeSH Terms: conditions — Skin Diseases; Keloid; Cicatrix; Fibrosis

STUDY DESIGN:
Intervention Model Description: Single-blind, dose escalation, randomized controlled Phase 1 study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HF-LED-RL Phototherapy (Experimental): The protocol for dose escalation requires subjects be enrolled sequentially in groups of five (three subjects randomized to HF-LED-RL phototherapy and two subjects randomized to mock therapy).
  After either a maximally tolerated dose (MTD) has been established or the study endpoint of 640 J/cm2 has been achieved, an additional 24 or 27 HF-LED-RL phototherapy subjects (for a total of 30) and 16 or 18 mock therapy subjects (for a total of 20) (determined randomly) will be enrolled to satisfy Hanley's Rule of Three, such that it can be concluded with 95% confidence that fewer than 1 person in 10 will experience an adverse event.
  Interventions: Device: HF-LED-RL Phototherapy
- Mock Therapy (Sham Comparator): The protocol for dose escalation requires subjects be enrolled sequentially in groups of five (three subjects randomized to HF-LED-RL phototherapy and two subjects randomized to mock therapy).
  After either a maximally tolerated dose (MTD) has been established or the study endpoint of 640 J/cm2 has been achieved, an additional 24 or 27 HF-LED-RL phototherapy subjects (for a total of 30) and 16 or 18 mock therapy subjects (for a total of 20) (determined randomly) will be enrolled to satisfy Hanley's Rule of Three, such that it can be concluded with 95% confidence that fewer than 1 person in 10 will experience an adverse event.
  Interventions: Device: Mock Therapy

INTERVENTIONS:
Device: HF-LED-RL Phototherapy — The starting dose of 480 J/cm2 will be administered to Group 1's HF-LED-RL phototherapy randomized subjects and the HF-LED-RL dose will be escalated in the subsequent group to 640 J/cm2. Common expected procedure side effects are mild and temporary, including warmth, redness (erythema) and swelling (edema). The maximally tolerated dose (MTD) is defined as the dose level below the dose producing unacceptable but reversible toxicity in 2 or more subjects and is considered the upper limit of subject tolerance.
  All subjects will receive total of nine LED-RL phototherapy, three times per week for three consecutive weeks.
  Other Names: Omnilux New-U (Photo Therapeutics, Carlsbad, CA)
  Arms: HF-LED-RL Phototherapy
Device: Mock Therapy — Mock therapy will be administered to mock therapy randomized subjects using the mock therapy unit. The mock therapy unit only generates warmth and does not emit LED-RL.
  All subjects will receive total of nine mock therapy procedures, three times per week for three consecutive weeks.
  Other Names: Mock therapy unit (Photo Therapeutics, Carlsbad, CA)
  Arms: Mock Therapy

SUMMARY:
The goal of this study is to establish the safety of high fluence LED-RL at fluence of 480 J/cm2 and 640 J/cm2 in healthy non-Hispanic, Caucasian subjects. The hypothesis is that high fluence LED-RL phototherapy is safe in non-Hispanic, Caucasians.

DETAILED DESCRIPTION:
The effects of visible light, while common in the environment (visible spectrum accounts for 44% of total solar energy), remain undefined. An important safety feature of visible red light (600 nm to 700 nm) is that it does not generate pro-carcinogenic DNA damage as does ultraviolet (UV) light. Recently published clinical observations indicate that red light in combination with other modalities such as photosensitizers in combined red light photodynamic therapy can treat skin diseases. However, preliminary in vitro data generated by the investigator's research group suggests that red light can function as a stand-alone treatment, eliminating the side-effects of chemical photosensitizers and the potential long-term harm of current UV therapy. Furthermore, commercially available light emitting diode-red light (LED-RL) units exist and are already FDA-cleared for other dermatological uses (such as rhytides and acne), thus clinical translation for use in skin diseases could occur relatively quickly following safety and efficacy demonstration. Developing high fluence LED-RL phototherapy as a treatment for skin conditions may represent an important advance that lacks the serious systemic side effects associated with immunomodulatory agents (such as oral steroids); avoids the need for invasive, painful injections with anti-fibrotic agents (such as intralesional steroids, 5-fluorouracil and bleomycin); and eliminates the UV-induced DNA damage associated with skin cancer and photoaging that are associated with current UVA/UVA1 and UVB/narrowband UVB phototherapy. To the investigator research group's knowledge, no clinical trials have been performed to determine the safety of high fluence LED-RL in different Fitzpatrick skin types. The innovation of this approach is that the investigator research group intend to study the safety of high fluence LED-RL in Fitzpatrick skin types I to III (based on NIH's race/ethnicity category of non-Hispanic, Caucasian).

A previous study demonstrated that fluence up to 320 J/cm2 is safe for all skin types (unpublished data, investigator research group). This study will evaluate doses of 480 J/cm2 and 640 J/cm2 in Fitzpatrick skin types I to III. This is based on the classical method for dose escalation as described by Spilker: starting with dose (X) increased by an equal amount (in this instance: X=160 J/cm2 which is the maximum recommended starting dose in clinical studies, 2X=320 J/cm2, 3X=480 J/cm2, 4X=640 J/cm2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of any sex and age
* Non-Hispanic, Caucasian race/ethnicity
* Nondominant proximal anterior forearm is wide enough to ensure reproducible placement of LED-RL phototherapy or mock therapy hand-held unit
* Available and willing to attend all clinic visits
* Able and willing to give informed consent

Exclusion Criteria:

* Subjects using any photosensitizers (i.e. lithium, melatonin, phenothiazine antipsychotics, antibiotics)
* Subjects with diabetes mellitus (DM)
* Subjects with a history of skin cancer.
* Subjects with systemic lupus erythematous (SLE)
* Subjects with light-sensitive conditions (All subjects will be tested for photosensitivity per manufacturer user guide instructions)
* Subjects with open wounds on the nondominant proximal anterior forearm
* Subjects with fibrotic skin disease or other skin conditions on the nondominant proximal anterior forearm
* Subjects with tattoos that cover the procedure site on the nondominant proximal anterior forearm
* Subjects of an ethnic race group other than Non-Hispanic, Caucasian
* Subjects who have previously participated in the VA Northern California's "Phase 1 Study of LED-RL in Human Skin"

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-01-08 (Estimated); Study Completion 2019-01-08 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 3 consecutive weeks
  The primary objective is to determine the maximum tolerated dose.

SECONDARY OUTCOMES:
Assessment of safety profile by evaluating incidence of procedure-related common procedure outcomes | 3 consecutive weeks
  To evaluate safety of high fluence LED-RL phototherapy by recording any common expected procedure outcomes [warmth, erythema (redness), and edema (swelling) that are mild, self-limited, and are expected to last less than 24 hours] via assessment during and immediately post-procedure and subject diary of adverse events.
Assessment of safety profile by evaluating incidence of adverse events | 3 consecutive weeks
  To evaluate safety of high fluence LED-RL phototherapy by recording adverse events (including: first-degree or higher skin burning or blistering, erythema lasting more than 24 hours, severe swelling, pain, ulceration, change in sensation, and/or muscle weakness], via assessment during and immediately post-procedure and subject diary of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD, MS, Principal Investigator — Physician, Dermatology
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jagdeo JR, Adams LE, Brody NI, Siegel DM. Transcranial red and near infrared light transmission in a cadaveric model. PLoS One. 2012;7(10):e47460. doi: 10.1371/journal.pone.0047460. Epub 2012 Oct 15. PMID 23077622
- [Background] Mamalis A, Jagdeo J. Light-emitting diode-generated red light inhibits keloid fibroblast proliferation. Dermatol Surg. 2015 Jan;41(1):35-9. doi: 10.1097/01.DSS.0000452650.06765.51. PMID 25485805
- [Background] Sadick NS. A study to determine the efficacy of a novel handheld light-emitting diode device in the treatment of photoaged skin. J Cosmet Dermatol. 2008 Dec;7(4):263-7. doi: 10.1111/j.1473-2165.2008.00404.x. PMID 19146602
- [Background] Sadick NS. Handheld LED array device in the treatment of acne vulgaris. J Drugs Dermatol. 2008 Apr;7(4):347-50. PMID 18459515
- [Background] Lev-Tov H, Mamalis A, Brody N, Siegel D, Jagdeo J. Inhibition of fibroblast proliferation in vitro using red light-emitting diodes. Dermatol Surg. 2013 Aug;39(8):1167-70. doi: 10.1111/dsu.12212. Epub 2013 Apr 16. PMID 23590233
- [Background] Ho D, Kraeva E, Wun T, Isseroff RR, Jagdeo J. A single-blind, dose escalation, phase I study of high-fluence light-emitting diode-red light (LED-RL) on human skin: study protocol for a randomized controlled trial. Trials. 2016 Aug 2;17:385. doi: 10.1186/s13063-016-1518-7. PMID 27484782
- [Derived] Wang EB, Kaur R, Nguyen J, Ho D, Austin E, Maverakis E, Li CS, Hwang ST, Isseroff RR, Jagdeo J. A single-blind, dose-escalation, phase I study of high-fluence light-emitting diode-red light on Caucasian non-Hispanic skin: study protocol for a randomized controlled trial. Trials. 2019 Mar 20;20(1):177. doi: 10.1186/s13063-019-3278-7. PMID 30894210

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT03433222/Prot_SAP_000.pdf